CLINICAL TRIAL: NCT00102362
Title: Job Seekers Training for Patients With Drug Dependence
Brief Title: Job-Seekers Training for Patients With Drug Dependence - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Maxine Stitzer, Ph.D., Johns Hopkins University
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized
Other Study IDs: NIDA-CTN-0020-1
Record Dates: First submitted 2005-01-27; First posted 2005-01-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to examine the effectiveness of a 12-hour basic job-training program designed to give drug abuse treatment patients the skills they need to find and secure a job and set vocational goals and methods for locating employment. The intervention to be evaluated is modeled after the Job Seekers' Workshop, which was manualized and has been tested in trials.

ELIGIBILITY:
* DSM-IV drug/alcohol abuse/dependence
* enrolled in drug treatment for at least 30 days
* unemployed or underemployed
* expressed interest in employment
* demonstrate English comprehension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627
Dates: Start 2004-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Employment or Job Training Program

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis, Ph.D., Principal Investigator — Johns Hopkins University
Locations (13):
- United States (13):
  - 14th Street Clinic, Berkely, California
  - Glenwood Life Counseling Center, Baltimore, Maryland
  - Man Alive, Baltimore, Maryland
  - Daybreak Rehabilitation Center, Baltimore, Maryland
  - CAB Health and Recovery Services, Inc., Danvers, Massachusetts
  - CAB Health Recovery-Salem Outpatient, Salem, Massachusetts
  - Psychiatry and Behavioral Medicine Professionals I, Detroit, Michigan
  - Self Help Addiction Rehabilitation (SHAR), Inc., Detroit, Michigan
  - Na'nizhoozhi Center, Inc., Gallup, New Mexico
  - Life Link, Santa Fe, New Mexico
  - New Directions, NW, Baker City, Oregon
  - Dorchester Alcohol and Drug Commission, Summerville, South Carolina
  - Chesterfield County CSB- Substance Abuse Services, Chesterfield, Virginia